CLINICAL TRIAL: NCT00495703
Title: Exercise Intervention for Chemotherapy-Related Cognitive Dysfunction
Brief Title: The Activity Intervention for Chemobrain
Acronym: TACTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Lance Armstrong Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: tactic
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Cancer; Chemotherapy; Cognitive Impairment
Keywords: Cancer survivors; Chemotherapy; Cognitive function; Exercise; Physical Activity
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Exercise
  Interventions: Behavioral: Exercise
- 2 (Active Comparator): Usual Care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Exercise — 6-months of regular aerobic exercise
  Arms: 1
Behavioral: Usual Care — 6-months of behavioral strategies to aid memory/cognition
  Arms: 2

SUMMARY:
Cognitive dysfunction following chemotherapy is an adverse treatment effect that impacts the quality of life for many cancer survivors receiving this adjuvant therapy. A strong body of evidence now indicates that that the initiation of a regular exercise program, at levels that are readily achievable by most adults (3-5 d/wk, 30-45 min/session), can improve cognitive function. Importantly, the domains of cognitive function that are enhanced by exercise participation are the same domains that are negatively affected by chemotherapy. Accordingly, we propose a 2 year research program that seeks to develop and test a safe, simple, and effective exercise intervention to optimize cognitive function following chemotherapy. To begin this research, we will: 1) conduct a randomized exercise intervention trial among cancer survivors that report persistent cognitive problems following chemotherapy (n=60), 2) explore possible mediators and moderators of the intervention on cognition in order to begin to understand how the intervention may work and for whom it may be most effective, and 3), conduct a cross-sectional study comparing cancer survivors enrolled in the trial (n=60) and matched controls (n=40) to evaluate the cognitive status among survivors in the intervention. We hypothesize that six-months of regular exercise will enhance cognitive function among cancer survivors, and that cancer survivors reporting cognitive dysfunction will have lower objectively measured cognitive performance than adults who have not received chemotherapy. To our knowledge this study would be the first to examine the influence of regular exercise participation on cognitive function among cancer survivors that experienced cognitive difficulties following chemotherapy.

DETAILED DESCRIPTION:
A substantial number of cancer survivors who receive chemotherapy report mild to moderate cognitive impairment following treatment. These impairments have been reported across a range of cancer types and chemotherapy agents. Adjuvant treatment has been reported to affect multiple cognitive domains, but three domains appear to be most strongly affected (i.e., executive functioning, declarative memory, motor function). Exercise participation, at levels that are readily achievable by most adults (3-5 d/wk, 30-45 min/d), preserves and enhances cognitive function. Importantly, domains that are enhanced by exercise overlap substantially with the domains adversely affected by chemotherapy. Accordingly, we propose a 2 year research program that seeks to develop and test a safe, simple, and effective exercise intervention to optimize cognitive function following chemotherapy. To begin this research, we will: 1) conduct a randomized exercise intervention trial among cancer survivors that report persistent cognitive problems following chemotherapy (exercise, n=30 vs. standard of care, n=30); 2) explore possible mediators and moderators of the intervention effect on cognition; and 3), conduct a cross-sectional study comparing cancer survivors enrolled in the trial (n=60) and matched controls (n=40) to evaluate the cognitive status among survivors in the intervention. We will employ a proven home-based exercise intervention and state of the art cognitive testing of relevant cognitive domains (e.g., Randt Memory Test, Trail Making B, Stroop task, T ask switching, Response compatibility) that we have used in preliminary studies. We hypothesize that six-months of regular exercise will enhance cognitive function among cancer survivors, and that cancer survivors reporting cognitive dysfunction will have lower objectively measured cognitive performance than adults who have not received chemotherapy. To our knowledge this study would be the first to examine the influence of regular exercise participation on cognitive function among cancer survivors that experienced cognitive difficulties following chemotherapy. Completion of this project will provide our research team with the necessary experience and intervention effectiveness information that will be used to conduct future more definitive trials.

ELIGIBILITY:
Inclusion Criteria:

- Non-metastatic cancer and received at least 4 cycles of chemotherapy, and report the onset of persistent cognitive difficulties following treatment Age 18+ yrs

Exclusion Criteria:

1. Have no prior diagnosis of cancer of the central nervous system,
2. Not have engaged in regular exercise in the past year (i.e., 5+ days/wk, 20+ min/d, 3+ months),
3. No cardiovascular disease or orthopedic problems that could be worsened by exercise as reported on the Physical Activity Readiness Questionnaire
4. No major systemic diseases (e.g., liver, kidney or adrenal diseases).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Objective measures of cognitive function (a test battery) | 6-months

SECONDARY OUTCOMES:
Exploratory analyses of psychological status, cardiorespiratory fitness, and inflammatory markers in blood. | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Charles E. Matthews, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States